CLINICAL TRIAL: NCT04086576
Title: Reducing Risky Drinking Using Smartphone Paired Breathalyzer
Brief Title: Breathalyzer Validation Study
Acronym: BVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 825273
Record Dates: First submitted 2019-09-03; First posted 2019-09-11 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Alcohol Drinking; Alcohol Intoxication
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Commercial Smartphone-paired breathalyzers-Set 1 (Experimental): All subjects will first be given a priming dose of alcohol containing vodka designed to raise the blood alcohol content based on weight and gender. Blood alcohol content will first be measured with three commercial smartphone-paired breathalyzers: Drivesafe Evoc, Alcohoot, and BacTrack Pro which will be tested in a randomized order and recorded. Participants blood alcohol content will also be measured using the Intoxilyzer 240, a police grade breathalyzer device After the tertiary dose of alcohol, a nurse will perform a blood draw on the participants, which will be used to determine blood alcohol content.
  Interventions: Device: Alcohoot; Device: BACtrack Mobile Pro; Device: DRIVESAFE Evoc; Device: Intoxilyzer 240
- Commercial Smartphone-paired breathalyzers-Set 2 (Experimental): All subjects will first be given a priming dose of alcohol containing vodka designed to raise the blood alcohol content based on weight and gender. Blood alcohol content will first be measured with three commercial smartphone-paired breathalyzers: BACtrack Vio, Drinkmate, and Floome which will be tested in a randomized order and recorded. Participants blood alcohol content will also be measured using the Intoxilyzer 240, a police grade breathalyzer device After the tertiary dose of alcohol, a nurse will perform a blood draw on the participants, which will be used to determine blood alcohol content.
  Interventions: Device: BACtrack Vio; Device: Drinkmate; Device: Floome; Device: Intoxilyzer 240

INTERVENTIONS:
Device: Alcohoot — Alcohoot branded smartphone-paired breathalyzer
  Arms: Commercial Smartphone-paired breathalyzers-Set 1
Device: BACtrack Mobile Pro — BACtrack Mobile Pro branded smartphone-paired breathalyzer
  Arms: Commercial Smartphone-paired breathalyzers-Set 1
Device: DRIVESAFE Evoc — DRIVESAFE Evoc branded smartphone-paired breathalyzer
  Arms: Commercial Smartphone-paired breathalyzers-Set 1
Device: BACtrack Vio — BACtrack Vio branded smartphone-paired breathalyzer
  Arms: Commercial Smartphone-paired breathalyzers-Set 2
Device: Drinkmate — Drinkmate branded smartphone-paired breathalyzer
  Arms: Commercial Smartphone-paired breathalyzers-Set 2
Device: Floome — Floome branded smartphone-paired breathalyzer
  Arms: Commercial Smartphone-paired breathalyzers-Set 2
Device: Intoxilyzer 240 — Intoxilyzer 240 police grade breathalyzer

SUMMARY:
The proposed project will test three commercial cellphone breathalyzers against a police grade breathalyzer device.The study will test the accuracy of these smartphone breathalyzers at assessing Breath Alcohol Content (BrAC) against a standard police grade breathalyzer. This study aims to fill the knowledge gap by determining the validity of smartphone paired breathalyzer devices to accurately assess BrAC. Data collection includes collection of BrAC measurements, as well as survey data.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-39 old
* Less than 4 drinking days and less than 12 drinks per week on average in the past 2 months
* Have previously consumed four (women) or five (men) or more standard drinks without problems
* A valid photo ID
* Willing to take public transportation home, via septa or an uber rideshare credit.

Exclusion Criteria:

* Desire alcohol treatment now or received it in the past 6 months
* Alcohol dependence with withdrawal per DSM-V criteria
* Non-English-speaking
* Individuals who have a medical condition or who are taking medication which limits or prevents the consumption of alcohol.

Ages: 21 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2017-04-17 (Actual); Study Completion 2017-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Kit Delgado, MD, MS, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alessi SM, Petry NM. A randomized study of cellphone technology to reinforce alcohol abstinence in the natural environment. Addiction. 2013 May;108(5):900-9. doi: 10.1111/add.12093. Epub 2013 Jan 30. PMID 23279560
- [Background] Easton CJ, Swan S, Sinha R. Prevalence of family violence in clients entering substance abuse treatment. J Subst Abuse Treat. 2000 Jan;18(1):23-8. doi: 10.1016/s0740-5472(99)00019-7. PMID 10636603
- [Background] Harrison EL, Fillmore MT. Are bad drivers more impaired by alcohol? Sober driving precision predicts impairment from alcohol in a simulated driving task. Accid Anal Prev. 2005 Sep;37(5):882-9. doi: 10.1016/j.aap.2005.04.005. PMID 15907777
- [Background] Harrison EL, Marczinski CA, Fillmore MT. Driver training conditions affect sensitivity to the impairing effects of alcohol on a simulated driving test [corrected]. Exp Clin Psychopharmacol. 2007 Dec;15(6):588-98. doi: 10.1037/1064-1297.15.6.588. PMID 18179312
- [Background] Kosten TR, O'Connor PG. Management of drug and alcohol withdrawal. N Engl J Med. 2003 May 1;348(18):1786-95. doi: 10.1056/NEJMra020617. No abstract available. PMID 12724485
- [Background] Loewenstein G, Brennan T, Volpp KG. Asymmetric paternalism to improve health behaviors. JAMA. 2007 Nov 28;298(20):2415-7. doi: 10.1001/jama.298.20.2415. No abstract available. PMID 18042920
- [Background] MacKillop J, Amlung MT, Few LR, Ray LA, Sweet LH, Munafo MR. Delayed reward discounting and addictive behavior: a meta-analysis. Psychopharmacology (Berl). 2011 Aug;216(3):305-21. doi: 10.1007/s00213-011-2229-0. Epub 2011 Mar 4. PMID 21373791
- [Background] Marczinski CA, Stamates AL. Artificial sweeteners versus regular mixers increase breath alcohol concentrations in male and female social drinkers. Alcohol Clin Exp Res. 2013 Apr;37(4):696-702. doi: 10.1111/acer.12039. Epub 2012 Dec 6. PMID 23216417
- [Background] McCarthy DM, Niculete ME, Treloar HR, Morris DH, Bartholow BD. Acute alcohol effects on impulsivity: associations with drinking and driving behavior. Addiction. 2012 Dec;107(12):2109-14. doi: 10.1111/j.1360-0443.2012.03974.x. Epub 2012 Aug 10. PMID 22690907
- [Background] McNeill JA, Sherwood GD, Starck PL, Thompson CJ. Assessing clinical outcomes: patient satisfaction with pain management. J Pain Symptom Manage. 1998 Jul;16(1):29-40. doi: 10.1016/s0885-3924(98)00034-7. PMID 9707655
- [Background] Patel MS, Asch DA, Volpp KG. Wearable devices as facilitators, not drivers, of health behavior change. JAMA. 2015 Feb 3;313(5):459-60. doi: 10.1001/jama.2014.14781. No abstract available. PMID 25569175
- [Background] Naimi TS, Brewer RD, Mokdad A, Denny C, Serdula MK, Marks JS. Binge drinking among US adults. JAMA. 2003 Jan 1;289(1):70-5. doi: 10.1001/jama.289.1.70. PMID 12503979
- [Background] Petry NM. A comprehensive guide to the application of contingency management procedures in clinical settings. Drug Alcohol Depend. 2000 Feb 1;58(1-2):9-25. doi: 10.1016/s0376-8716(99)00071-x. PMID 10669051
- [Background] Petry NM, Martin B, Cooney JL, Kranzler HR. Give them prizes, and they will come: contingency management for treatment of alcohol dependence. J Consult Clin Psychol. 2000 Apr;68(2):250-7. doi: 10.1037//0022-006x.68.2.250. PMID 10780125
- [Background] Prendergast M, Podus D, Finney J, Greenwell L, Roll J. Contingency management for treatment of substance use disorders: a meta-analysis. Addiction. 2006 Nov;101(11):1546-60. doi: 10.1111/j.1360-0443.2006.01581.x. PMID 17034434
- [Background] Roll JM, Petry NM, Stitzer ML, Brecht ML, Peirce JM, McCann MJ, Blaine J, MacDonald M, DiMaria J, Lucero L, Kellogg S. Contingency management for the treatment of methamphetamine use disorders. Am J Psychiatry. 2006 Nov;163(11):1993-9. doi: 10.1176/ajp.2006.163.11.1993. PMID 17074952
- [Background] Senecal N, Wang T, Thompson E, Kable JW. Normative arguments from experts and peers reduce delay discounting. Judgm Decis Mak. 2012 Sep 1;7(5):568-589. PMID 23596504
- [Background] Sloan FA, Eldred LM, Xu Y. The behavioral economics of drunk driving. J Health Econ. 2014 May;35:64-81. doi: 10.1016/j.jhealeco.2014.01.005. Epub 2014 Feb 11. PMID 24603444
- [Background] Van Dyke N, Fillmore MT. Acute effects of alcohol on inhibitory control and simulated driving in DUI offenders. J Safety Res. 2014 Jun;49:5-11. doi: 10.1016/j.jsr.2014.02.004. Epub 2014 Mar 22. PMID 24913486
- [Background] Watson PE, Watson ID, Batt RD. Prediction of blood alcohol concentrations in human subjects. Updating the Widmark Equation. J Stud Alcohol. 1981 Jul;42(7):547-56. doi: 10.15288/jsa.1981.42.547. No abstract available. PMID 7289599
- [Background] White A, Hingson R. The burden of alcohol use: excessive alcohol consumption and related consequences among college students. Alcohol Res. 2013;35(2):201-18. doi: 10.35946/arcr.v35.2.11. PMID 24881329

RESULTS

PARTICIPANT FLOW:
Groups:
- Commercial Smartphone-paired Breathalyzers-Set 1: Smartphone-paired mobile breathalyzer-Set 1: All subjects will first be given a priming dose of alcohol containing vodka designed to raise the blood alcohol content based on weight and gender. Blood alcohol content will first be measured with three commercial smartphone-paired breathalyzers: Drivesafe Evoc, Alcohoot, and BacTrack Pro which will be tested in a randomized order and recorded. Participants' blood alcohol content will also be measured using the Intoxilyzer 240, a police grade breathalyzer device. After the tertiary dose of alcohol, a nurse will perform a blood draw on the participants, which will be used to determine blood alcohol content.
- Commercial Smartphone-paired Breathalyzers-Set 2: Smartphone-paired mobile breathalyzer-Set 2: All subjects will first be given a priming dose of alcohol containing vodka designed to raise the blood alcohol content based on weight and gender. Blood alcohol content will first be measured with three commercial smartphone-paired breathalyzers: BACtrack Vio, Drinkmate, and Floome which will be tested in a randomized order and recorded. Participants' blood alcohol content will also be measured using the Intoxilyzer 240, a police grade breathalyzer device. After the tertiary dose of alcohol, a nurse will perform a blood draw on the participants, which will be used to determine blood alcohol content.
Period: Overall Study
Arm/Group | Commercial Smartphone-paired Breathalyzers-Set 1 | Commercial Smartphone-paired Breathalyzers-Set 2
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Commercial Smartphone-paired Breathalyzers-Set 1 | Commercial Smartphone-paired Breathalyzers-Set 2 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (3.9) | 26.3 (2.5) | 26.8 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI (mean ± SD) [Mean (Standard Deviation); unit: kg/m^2] | 24.4 (4.6) | 24.7 (4.3) | 24.6 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Alcohol in Breath Variability
Description: Difference in Breath Alcohol Concentration (BrAC) from police-grade (Intoxilyzer 240) and consumer smartphone-paired breath testing devices relative to Blood Alcohol Concentration (BAC) measured from blood draw after tertiary dose of alcohol.
Time Frame: 8 Hours
Population: Group 1: Alcohoot, Evoc, BACtrack Mobile Pro, Intoxilyzer 240 (A). Group 2: BACtrack Vio, Drinkmate, Floome, Intoxilyzer 240 (B). Percent of Alcohol in Blood - grouped.
Measure: Mean (Standard Deviation); unit: percentage of alcohol
Groups:
- Intoxilyzer 240 (A); Intoxilyzer 240 (B): Intoxilyzer 240 police grade breathalyzer
- Drinkmate: Drinkmate branded smartphone-paired breathlyzer
- Percent of Alcohol in Blood: Percentage of Alcohol in Blood measured from blood draw
Arm/Group | Alcohoot | BACtrack Mobile Pro | DRIVESAFE Evoc | Intoxilyzer 240 (A) | BACtrack Vio | Drinkmate | Floome | Intoxilyzer 240 (B) | Percent of Alcohol in Blood
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 20
percentage of alcohol | 0.0912 (0.0164) | 0.0968 (0.0147) | 0.0694 (0.0074) | 0.0912 (0.0099) | 0.0746 (0.0312) | 0.0495 (0.0181) | 0.0770 (0.0194) | 0.0860 (0.0160) | 0.0996 (0.0165)
Statistical Analysis 1: Comparison: Intoxilyzer 240 (A) vs Intoxilyzer 240 (B); Each breathalyzer is compared to the percentage of alcohol in the blood during the time of blood draw (90 minutes); Test type: Superiority; p < .0001, ANOVA — Yes, used Tukey Kramer pairwise comparisons to adjust for multiple comparisons; ANOVA in repeated measures

2. Secondary Outcome: Differences in Readings on Devices for Percentage of Alcohol in Breath
Description: Mean difference in percent of blood in breath (BrAC) between the police-grade and personal, commercial breath testing devices
Time Frame: 8 Hours
Measure: Mean (95% Confidence Interval); unit: percentage of alcohol in breath
Arm/Group | Alcohoot | BACtrack Mobile Pro | DRIVESAFE Evoc | BACtrack Vio | Drinkmate | Floome
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
percentage of alcohol in breath | -0.000836 [-0.003066 to 0.001394] | 0.005853 [0.003643 to 0.008064] | -0.015698 [-0.017905 to -0.013491] | -0.000405 [-0.00345 to 0.002639] | -0.014616 [-0.017642 to -0.01159] | -0.006004 [-0.009094 to -0.002915]

ADVERSE EVENTS:
Time Frame: 8 hours
Description: Screening for eligibility reduced risk of all risk mortality
Arm/Group | Commercial Smartphone-paired Breathalyzers-Set 1 | Commercial Smartphone-paired Breathalyzers-Set 2
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT04086576/Prot_SAP_000.pdf